CLINICAL TRIAL: NCT03462511
Title: Hydroxyurea Adherence for Personal Best in Sickle Cell Disease (HABIT): Efficacy Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Arlene Smaldone, Professor of Nursing, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAR2908; 1R01NR017206-01 (NIH)
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Sickle Cell Disease
Keywords: Hydroxyurea; Community health worker (CHW); Text messages; Medication adherence
MeSH Terms: conditions — Anemia, Sickle Cell; Medication Adherence | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Dyads randomized to the control group will receive:
  Standard care and Education handouts.
  Interventions: Other: Standard of Care; Other: Education materials
- Intervention Group (Experimental): In addition to standard care and education handouts, dyads randomized to the intervention group will receive the HABIT intervention, which includes CHW support and tailored text messages.
  Interventions: Behavioral: HABIT Intervention; Other: Standard of Care; Other: Education materials

INTERVENTIONS:
Behavioral: HABIT Intervention — Dyads randomized to the intervention group will receive the HABIT intervention, which includes CHW support and tailored text messages.
  Arms: Intervention Group
Other: Standard of Care — Standard of care used to treat patients with SCD
Other: Education materials — Education materials provided to all patients enrolled in the trial

SUMMARY:
Many youth with chronic disease have difficulty taking medication every day and therefore do not receive full benefit from treatment. Sickle Cell Disease (SCD) is an inherited blood disease that affects African Americans and other underserved communities. Hydroxyurea (HU) is the sole FDA-approved drug therapy for SCD and is highly effective and improves quality of life. The proposed study, a 5-site four-year randomized control trial (RCT), builds upon the investigators' recent feasibility study of the same title. Overall goals are reducing barriers to HU use and improving adherence for youth 10-18 years through creation of a daily medication habit. The goal of the proposed multi-site study is to test the efficacy of the HABIT intervention at 6 months and sustainability of the effect at 12 months.

DETAILED DESCRIPTION:
Barriers to medication adherence are common in youth with chronic illness and are a source of racial/ethnic disparities in underserved communities. An inherited blood disease, Sickle Cell Disease (SCD) is characterized by chronic and acute illness and reduced quality of life (QOL). It affects African Americans and other underserved communities. Hydroxyurea (HU) is the sole FDA-approved drug therapy for SCD and is highly effective and improves QOL. Poor adherence is common among youth and young adults with SCD.

The importance of poor medication adherence, use of community-based health workers (CHWs) to bridge the gap between health services and underserved parent-youth dyads affected by SCD, the strength of the science, the success of the investigators' multi-ethnic feasibility study, and the potential application of study findings to youth with other serious chronic illnesses speak to the importance of this trial.

ELIGIBILITY:
Inclusion Criteria - Youth:

* One of the two most common sickle cell disease variants (HbSS or HbS-B0 thalassemia)
* Age 10 through18 years (inclusive)
* Currently prescribed hydroxyurea (HU) ≥18 months (for identifying historical Personal best HbF)
* Current HU dose is within 5% of dose at Personal Best HbF
* Pre-enrollment HbF ≥15% below historical Personal best, based on mean of ≥2 HbF assessments over preceding 12 months
* Youth able to speak/read English or Spanish

Inclusion Criteria - Parent:

* Parent/guardian speaks/reads English or Spanish
* Parent/ legal guardian willing to participate
* Family expects to reside in community for ≥ 1.5 years

Exclusion Criteria - Youth:

* Youth not prescribed HU
* <2 HbF assessments over past 12 months
* Transfusion within 3 months preceding enrollment
* Final screen HbF (visit 0) of ≤15% decrease below Personal best HbF
* Sexually active female 10 years or older and not using reliable contraception (due to HU teratogenic risk)
* Pregnancy
* Cognitive impairment (>2 levels below expected grade)
* Youth not residing with parent/legal guardian

Exclusion Criteria - Parent:

* Parent/legal guardian does not reside with youth

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Smaldone, PhD, CPNP-PC, Principal Investigator — Columbia University School of Nursing; Nancy S Green, MD, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - Feinstein Institute for Medical Research, Manhasset, New York
  - Columbia University Irving Medical Center, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruzzese JM, Usseglio J, Iannacci-Manasia L, Diggs KA, Smaldone AM, Green NS. Mental and Emotional Health of Caregivers of Youth with Sickle Cell Disease: A Systematic Review. J Health Care Poor Underserved. 2023;34(3):1070-1104. PMID 38015138
- [Background] Askew MA, Smaldone AM, Gold MA, Smith-Whitley K, Strouse JJ, Jin Z, Green NS. Pediatric hematology providers' contraceptive practices for female adolescents and young adults with sickle cell disease: A national survey. Pediatr Blood Cancer. 2022 Oct;69(10):e29877. doi: 10.1002/pbc.29877. Epub 2022 Jul 20. PMID 35856776
- [Background] Smaldone A, Manwani D, Aygun B, Smith-Whitley K, Jia H, Bruzzese JM, Findley S, Massei J, Green NS. HABIT efficacy and sustainability trial, a multi-center randomized controlled trial to improve hydroxyurea adherence in youth with sickle cell disease: a study protocol. BMC Pediatr. 2019 Oct 15;19(1):354. doi: 10.1186/s12887-019-1746-6. PMID 31615480
- [Result] Green NS, Manwani D, Aygun B, Appiah-Kubi A, Smith-Whitley K, Castillo Y, Soriano L, Jia H, Smaldone AM. Hydroxyurea Adherence for Personal Best in Sickle Cell Treatment (HABIT) efficacy trial: Community health worker support may increase hydroxyurea adherence of youth with sickle cell disease. Pediatr Blood Cancer. 2024 Apr;71(4):e30878. doi: 10.1002/pbc.30878. Epub 2024 Feb 6. PMID 38321562
- [Result] Green NS, Manwani D, Smith-Whitley K, Aygun B, Appiah-Kubi A, Smaldone AM. Mental health assessment of youth with sickle cell disease and their primary caregivers during the COVID-19 pandemic. Pediatr Blood Cancer. 2022 Sep;69(9):e29797. doi: 10.1002/pbc.29797. Epub 2022 May 25. PMID 35614571
- [Derived] Lalji R, Koh L, Francis A, Khalid R, Guha C, Johnson DW, Wong G. Patient navigator programmes for children and adolescents with chronic diseases. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD014688. doi: 10.1002/14651858.CD014688.pub2. PMID 39382077

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 24 Dyads were randomized to the intervention (24 parents + 24 youth) 26 Dyads were randomized to the control (26 parents + 26 youth)
Groups:
- Intervention Group: In addition to standard care and education handouts, dyads randomized to the intervention group will receive the HABIT intervention, which includes community health workers (CHW) support and tailored text messages.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 24 (24 Dyads (48 Unique individuals: 24 parents + 24 youth)) | 26 (26 Dyads (52 Unique Individuals: 26 parents + 26 youth))
Completed | 22 (22 Dyads (44 Unique Individuals: 22 Parents + 22 youth)) | 23 (23 Dyads (46 Unique Individuals: 23 Parents + 23 Youth))
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Population: The following variables were collected for children: Age, Sex, Race, Ethnicity, No other chronic conditions besides sickle cell disease, Number of emergency room visits, Number of hospitalizations, Biomarker fetal hemoglobin, Proportion of days covered by hydroxyurea The following variables were collected for parent/primary caregiver: Parent status, Parent education, Caregiver affected by sickle cell disease, Other people at home affected by sickle cell disease
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (1.9) | 13.0 (1.7) | 13.3 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 12 | 15 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 21 | 21 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 20 | 41
  White | 0 | 0 | 0
  More than one race | 3 | 6 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 50
No other chronic condition besides Sickle Cell Disease (SCD) [Count of Participants; unit: Participants] | 12 | 13 | 25
Had 1 or more ED visits in past year [Count of Participants; unit: Participants] — Participants with one or more emergency department (ED) visits in the year prior to enrollment
  Participants | 11 | 10 | 21
Had 1 more hospitalizations in past year [Count of Participants; unit: Participants] — Participants with one or more hospitalizations in the year prior to enrollment
  Participants | 11 | 11 | 22
Parent status: Single, separated or divorced [Count of Participants; unit: Participants] | 16 | 16 | 32
Parent education high school or less [Count of Participants; unit: Participants] | 7 | 14 | 21
Caregiver affected by SCD [Count of Participants; unit: Participants] | 2 | 1 | 3
Other people in home affected by SCD [Count of Participants; unit: Participants] | 4 | 6 | 10
Biomarker Fetal Hemoglobin (HbF) [Mean (Standard Deviation); unit: Percent] — Measure of the percentage of fetal hemoglobin in the blood
  Percent | 12.2 (5.9) | 12.4 (5.3) | 12.3 (5.5)
Proportion of days covered by hydroxyurea [Mean (Standard Deviation); unit: Percent of days] — The proportion of days covered by hydroxyurea in the year prior to study enrollment, using prescription refill data.
  Percent of days | 55.2 (26.7) | 55.9 (26.1) | 55.6 (26.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Biomarker Fetal Hemoglobin (HbF)
Description: A serum biomarker obtained from youth used to measure adherence to hydroxyurea
Time Frame: Baseline, 6 months, 12 months
Population: Change between 6-12 months: 22 of 24 intervention group participants analyzed as blood samples were collected at both timepoints for 22 of 24 participants, due to difficulties coming into clinic during the COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: Percent fetal hemoglobin
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 24 | 26
Percent fetal hemoglobin
  Baseline to Month 6 | 2.7 (1.3) | 0.3 (1.3)
  Month 6 to Month 12: number analyzed (Participants) | 22 | 26
  Month 6 to Month 12 | -1.7 (1.2) | 1.8 (1.3)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Based on estimated effect size from our prior feasibility trial, the target enrollment was 87 dyads plus additional 20% to account for attrition before Month 6 or blood transfusions or acute illness rendering HbF levels inaccurate; Test type: Superiority; p = 0.067, Regression, Linear — Independent variables: study month, study group, their interactions and a person-level random intercept to incorporate clustering; Mean Difference (Net) = 2.4

2. Primary Outcome: Mean Change in Proportion of Days Covered (PDC) by Hydroxyurea
Description: The days covered by hydroxyurea was assessed using youth prescription refill data and was used to measure hydroxyurea adherence. The baseline measure is the proportion of days covered by hydroxyurea in the year prior to study enrollment, using prescription refill data.
Time Frame: Baseline, 6 months, 12 months
Population: 21 of 24 intervention group participants and 22 of 26 control group participants analyzed as data could not be collected from pharmacies due to COVID-19 difficulties and loss of data resulting from fire.
Measure: Mean (Standard Deviation); unit: change in percentage of PDC
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 21 | 22
change in percentage of PDC
  Baseline and 6 months | 17.9 (27.3) | 13.1 (29.7)
  6 months and 12 months | -1.6 (22.8) | -1.9 (33.7)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; We compared the difference in proportion of days covered by hydroxyurea at two timepoints: (1) from the year prior to study entry to 6 months (the end of the active intervention phase of the trial) and (2) from 6 months to 12 months (the sustainability phase of the trial); Test type: Superiority; p = 0.60, t-test, 2 sided

3. Secondary Outcome: Mean Change in Youth Score on Peds Quality of Life (Generic Quality of Life)
Description: Used to measure health-related quality of life. Scores range from 0-100 with a higher score indicating a better quality of life.
Time Frame: Baseline, 4 months, 9 months and 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 24 | 26
score on a scale
  Baseline to 9 months | 10.3 (12.6) | 2.0 (12.3)
  9 months to 12 months | -2.5 (11.6) | 1.1 (16.2)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; We hypothesized that, compared to the control group, generic quality of life (QOL) for youth in the intervention group would improve from baseline to 9 months; Test type: Superiority; p < 0.001, Regression, Linear
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; We hypothesized that the improvement in quality of life experienced by the intervention group would be sustained from month 9 to month 12; Test type: Non-Inferiority — 30% of the standard deviation was used as the non-inferiority margin. For this test generic quality of life (QOL) scores for months 4-9 (efficacy period) were compared to months >9 (sustainability period); p = 0.04, Regression, Linear

4. Secondary Outcome: Mean Change in Youth Score on PedsQL Sickle Cell Disease Module (Disease Specific Quality of Life)
Description: Used to measure sickle cell disease specific health-related quality of life. Scores range from 0-100 with a higher score indicating a better quality of life.
Time Frame: Baseline, 9 months and 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 24 | 26
score on a scale
  Baseline to 9 months | 16.4 (23.3) | 9.0 (12.0)
  9 months to 12 months | -4.3 (21.9) | -0.7 (15.7)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; We hypothesized that, compared to the control group, sickle cell disease specific quality of life (SC-QOL) for youth in the intervention group would improve from baseline to 9 months; Test type: Superiority; p = 0.47, Regression, Linear
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; We hypothesized that the improvement in sickle cell disease specific quality of life (SC-QOL) experienced by the intervention group would be sustained from month 9 to month 12; Test type: Non-Inferiority — 30% of the standard deviation was used as the non-inferiority margin. For this test sickle cell disease specific quality of life (SC-QOL) scores for months 4-9 (efficacy period) were compared to months >9 (sustainability period); p = 0.045, Regression, Linear

5. Secondary Outcome: Mean Change in Parent Youth Concordance Regarding Self-management Responsibility
Description: Concordance between parent and youth scores Sickle Cell Family Responsibility scores for 11 items measuring self-management tasks. Scores range from 0-11 with a higher score indicating better concordance.
Time Frame: Baseline, 6 months and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 24 | 26
units on a scale
  Baseline to 6 months | 1.6 (2.4) | 1.4 (2.5)
  6 months to 12 months | 0.3 (2.1) | 0.5 (2.3)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; We hypothesized that, compared to the control group, responsibility for self-management concordance for youth-caregiver dyads in the intervention group would improve from baseline to 6 months; Test type: Superiority; p = 0.002, Regression, Linear
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; We hypothesized that the improvement in concordance between youth and caregivers for self-management responsibility experienced by the intervention group would be sustained from month 6 to month 12; Test type: Non-Inferiority — 50% of the standard deviation was used as the non-inferiority margin. For this test youth caregiver concordance for self-management responsibility scores for months 0-6 (efficacy period) were compared to months 6-12 (sustainability period); p = 0.23, Regression, Linear

ADVERSE EVENTS:
Time Frame: 12 months
Description: AE data were only collected on youth
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT03462511/Prot_SAP_000.pdf